CLINICAL TRIAL: NCT05077501
Title: A Prospective, Phase I, Double-blind, Parallel-group, Placebo-controlled, Randomised Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Oral Doses of ACD856 in Healthy Volunteers
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of ACD856
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AlzeCure Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2000CI-002
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease; Cognition Disorder
Keywords: Alzheimer's Disease; Cognition Disorder
MeSH Terms: conditions — Alzheimer Disease; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACD856 (Experimental)
  Interventions: Drug: ACD856
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACD856 — Multiple daily oral doses of ACD856 will be administered for 7 days in an escalation scheme of dose 1, dose 2 and dose 3. The escalation schedule may be adapted based on evaluation by the internal Safety Review Committee.
  Arms: ACD856
Drug: Placebo — Placebo oral solution
  Arms: Placebo

SUMMARY:
The multiple ascending dose (MAD) design of the study is based on the aim to study safety, tolerability, PK and pharmacodynamics of selected doses of ACD856 in a limited number of healthy volunteers.

ACD856 will be administered orally.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to any study-mandated procedure.
* Willing and able to comply with study requirements.
* Healthy male or female adults of non-childbearing potential aged ≥ 18 and ≤ 65 years at screening.
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 at screening.
* Only subjects of non-childbearing potential may be included in the study. Male subjects with partners of childbearing potential must be willing to use condoms, be vasectomised or practice sexual abstinence to prevent pregnancy and drug exposure of a partner, as well as refrain from donating sperm from the date of dosing until 3 months after dosing with the IMP.
* Clinically acceptable medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.

Exclusion Criteria:

* Any exposure to ACD856 in the past.
* Treatment with another investigational drug within 3 months prior to or during the study.
* Positive screen for drugs of abuse or a positive alcohol result at screening or admission to the clinic.
* Clinically relevant findings in laboratory parameters, ECG or vital signs at screening.
* Current smokers or subjects who use nicotine products.
* History of alcohol abuse or excessive intake of alcohol.
* History of, or current use of, anabolic steroids.
* Excessive caffeine consumption.
* Plasma donation or blood donation prior to screening.
* Any planned night shift work within the duration of the study, from 48 h prior to randomisation until follow-up.
* Any planned major surgery within the duration of the study.
* Evidence of an active infection that requires treatment with antibiotics within 2 weeks of planned dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) | 16 days
  Number and percentage of subjects with adverse events (AEs).
Clinically significant changes in 12-lead ECGs | 16 days
  Number of subjects and percentage of subjects with clinically significant changes in 12-lead ECGs
Clinically significant changes in vital signs | 16 days
  Number of subjects and percentage of subjects with clinically significant changes in vital signs or stool frequency
Clinically significant changes in hematology, clinical chemistry, coagulation and/or urinalysis parameters | 16 days
  Number of subjects and percentage of subjects with clinically significant changes in any safety laboratory assessments.
Clinically significant changes in physical examinations | 16 days
  Number of subjects and percentage of subjects with clinically significant changes in physical examinations
GAD-7 | 16 days
  Change from baseline of GAD-7
PHQ-9 | 16 days
  Change from baseline of PHQ-9
C-SSRS | 16 days
  Change from baseline of C-SSRS
Prolactin | 10 days
  Change from baseline of prolactin levels

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sandin, PhD, Study Director — AlzeCure Pharma
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No